CLINICAL TRIAL: NCT07199803
Title: Comparing the Obstetric Quality of Recovery-10 (OBS-QoR-10) in Patients With and Without Postpartum Hemorrhage: A Matched Case-control Study
Brief Title: OBS-QoR-10 in Patients With and Without Postpartum Hemorrhage
Status: Recruiting | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 25-03
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Postpartum Hemorrhage (Primary)
Keywords: cesarean delivery; vaginal delivery; ObsQoR-10
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Vaginal delivery with PPH: Patients who deliver vaginally with a quantitative blood loss greater than or equal to 1000ml.
  Interventions: Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool
- Vaginal delivery without PPH: Patients who deliver vaginally with a quantitative blood loss less than 1000ml.
  Interventions: Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool
- Cesarean delivery with PPH: Patients who deliver vaginally with a quantitative blood loss greater than or equal to 1000ml.
  Interventions: Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool
- Cesarean delivery without PPH: Patients who deliver vaginally with a quantitative blood loss less than 1000ml.
  Interventions: Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool

INTERVENTIONS:
Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool — The ObsQoR-10 tool aims to quantitatively measure functional recovery at 24 hours postpartum. It includes 10 questions on a 0 to 10 scale, aimed at pain management, the adverse effects of narcotics and the perception of recovery by the patient.

SUMMARY:
Postpartum hemorrhage (PPH) remains a leading cause of maternal death and morbidity. Moreover, it also contributes to psychological trauma such as depression and post-traumatic stress disorder. The American College of Obstetrics and Gynecology (ACOG) and the Society for Maternal Fetal Medicine (SMFM) defines this morbidity as an unintended outcome in the birthing process that may have significant short-term and long-term consequences to an individual's health. A recent study in 2018 developed core outcomes set for PPH through Delphi consensus encompassing elements of prevention and management of PPH.

Patient-reported outcomes, breastfeeding, and overall sense of wellbeing were not included in the final outcome set. Nevertheless, investigators felt strongly that they should be included, but further work was needed to assess the factors influencing the quality of recovery in the context of PPH. This is aligned with increasing recognition that patient experiences are important to improving the quality of care and quality of recovery after Cesarean delivery. The most effective, i.e. validated tool for assessing postpartum recovery is the Obstetric Quality of Recovery-10 (Obs-QoR-10). However its application in patients with PPH remains unexplored. It would appear logical that patient experiencing PPH experience a potentially more challenging recovery process which may include more surgical complications, depressive symptoms, sleep deprivation, physical exhaustion and stress due to unexpected and undesired delivery events. This study aims to compare Obs-QoR-10 scores in patients with and without PPH to evaluate the impact of severe postpartum bleeding on recovery outcomes using a matched case-control design.

The investigators plan to determine the differences in Obs-QoR-10 scores between patients who experience PPH during childbirth and those deliver without PPH, and to evaluate the impact of PPH on specific recovery domains (physical comfort, emotional well-being, and functional recovery).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who have delivered at Mount Sinai Hospital.
* Delivery via vaginal or cesarean delivery with neuraxial analgesia or anesthesia
* Ability to communicate in English (to answer OBSQoR-10 survey) PPH Cohort

  * Quantitative Blood Loss (QBL) ≥ 1000 mL or,
  * Transfusion of blood due to PPH or,
  * Transfer to ICU level care due to PPH
  * Significant PPH intervention, i.e. hysterectomy or arterial embolization Non-PPH
  * QBL < 500 mL and,
  * No transfusion of blood products, and
  * No need for elevated care environment, i.e. HAU or ICU

Exclusion Criteria:

* Patients with pre-existing psychiatric disorders affecting recovery assessment.
* Patients who experience severe obstetric complications other than PPH (e.g., eclampsia, uterine rupture).
* Overdistended uterus due to; Polyhydramnios (amniotic fluid index >24 cm) or multiple gestation
* History of previous PPH (documented with blood loss of >1000 ml, blood transfusion, use surgical methods such as Bakri balloon, B-Lynch sutures, uterine artery ligation or embolization)
* BMI > 50
* Language barrier (English)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that deliver at Mount Sinai Hospital with measured blood loss greater than or equal to 1000ml, and a set of controls matching the following criteria with measured blood loss less than 1000ml:
  * Age (±5 years)
  * Parity (1 or >1)
  * Mode of delivery (vaginal vs. cesarean delivery)
  * Labour (Labouring and Non-labouring cesarean delivery)
  * Urgency (Scheduled vs Unscheduled Cesarean delivery)
  * Gestational age at delivery (± 2 weeks)
  * Delivery date within 2 weeks
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2025-10-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) score 24-48 hours | 24 hours
  ObsQoR-10 score between 24 and 48 hours postpartum. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.

SECONDARY OUTCOMES:
Semi-quantitative blood loss total (ml) | 1 hour
  Semi-quantitative blood loss total (ml) as measured postpartum
Length of hospital stay (hours) | 4 days
  Time from admission to discharge from hospital in hours
Additional uterotonic medication administered - questionnaire | 24 hours
  Presence of administration and dosing of any additional uterotonic medication.
Blood transfusion | 48 hours
  Administration of any blood product and amount given.
Surgical interventions for PPH - questionnaire | 2 hours
  Use of any surgical interventions for PPH as documented by the surgical team.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald George, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No